CLINICAL TRIAL: NCT07277660
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Galvokimig in Adult Study Participants With Moderate to Severe Atopic Dermatitis
Brief Title: A Dose-ranging Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Galvokimig in Adult Study Participants With Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATD002; 2025-522578-35 (Registry Identifier: CTIS (EU)); U1111-1326-9886 (Other: Universal Trial Number (UTN))
Record Dates: First submitted 2025-12-02; First posted 2025-12-11 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Galvokimig,; UCB9741
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Galvokimig Arm 1 (Experimental): Participants will receive a predefined Galvokimig Dose during Initial Intervention Period. After week 16 participants will continue on the same or a modfied dose.
  Interventions: Biological: Galvokimig
- Galvokimig Arm 2 (Experimental): Participants will receive a predefined Galvokimig Dose during Initial Intervention Period. After week 16 participants will continue on the same or a modfied dose.
  Interventions: Biological: Galvokimig
- Galvokimig Arm 3 (Experimental): Participants will receive a predefined Galvokimig Dose during Initial Intervention Period. After week 16 participants will continue on the same or a modfied dose.
  Interventions: Biological: Galvokimig
- Placebo (Placebo Comparator): Participants will receive matching placebo during Initial Intervention Period. After week 16 participants will continue on the same or a dose galvokimig.
  Interventions: Biological: Galvokimig; Drug: Placebo

INTERVENTIONS:
Biological: Galvokimig — Drug: Galvokimig Pharmaceutical form: Solution for injection
  Other Names: UCB9741
Drug: Placebo — Drug: Placebo Pharmaceutical form: Solution for injection
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the dose-response relationship of galvokimig compared with placebo in study participants with moderate-to-severe atopic dermatitis (AtD).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be aged greater than or equal (≥)18 years at the time of signing the informed consent
* Participant has chronic atopic dermatitis (AtD) (according to American Academy of Dermatology Consensus Criteria) that has been present for at least ≥1 year prior to initiating the study (ie, signing of the informed consent form [ICF]) and with:

  1. validated Investigator Global Assessment (vIGA) score ≥3 at Screening and Baseline
  2. Eczema Area and Severity Index (EASI) score ≥16 at both Screening and Baseline
  3. Peak Pruritus Numerical Rating Scale (PP-NRS) score of ≥4 at both Screening and Baseline
  4. ≥10% body surface area (BSA) of AtD involvement at both Screening and Baseline
  5. Documented recent history (within 6 months prior to Screening) of inadequate response to treatment with topical medications, or study participants for whom topical treatments are otherwise medically inadvisable (eg, due to important side effects or safety risks) and who are candidates for systemic therapy

Exclusion Criteria:

* Participant has any history or presence of any medical or psychiatric condition, physical examination finding, laboratory test result, or electrocardiogram (ECG) signal that, in the opinion of the investigator, could constitute a risk when taking the study intervention; or interfere with the interpretation of data and could jeopardize or would compromise the study participant's ability to participate in this study
* Active dermatologic conditions that may confound the diagnosis of AtD or would interfere with assessment of treatment, such as but not limited to scabies, seborrheic dermatitis, cutaneous lymphoma, ichthyosis, psoriasis, active allergic or irritant contact dermatitis
* Presence or family history (first degree) of inflammatory bowel disease (includes Crohn's disease and ulcerative colitis)
* History of chronic or recurrent infections, or a serious or life-threatening infection within the 6 months prior to the Baseline (including herpes zoster) as judged by the investigator
* Participants are not permitted to enroll into the study if they meet tuberculosis (TB) exclusion criteria
* Previous treatment with galvokimig
* Participant has relevant safety events to one or more interleukin (IL)-13 biologic response modifiers (ie, dupilumab, tralokinumab and lebrikizumab) that resulted in discontinuation and change of treatment
* All systemic therapies (other than biologics), topical therapies and other treatments for AtD must be discontinued at least 4 weeks prior to Baseline
* Treatment with biologic agents must discontinued at least 3 months prior to baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2027-05-17 (Estimated); Study Completion 2028-03-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with Eczema Area and Severity Index (EASI)75 response at Week 16 | Week 16
  The EASI is a validated scoring system that grades the physical signs of atopic dermatitis/eczema.
  The severity of each clinical sign is scored as: 0=None to 3=Severe.

SECONDARY OUTCOMES:
Percentage of Participants with validated Investigator Global Assessment (vIGA) response at Week 16 | Week 16
  The vIGA score is using descriptors that best describe the overall appearance of the lesions at a given time point. Assessment: vIGA 0=clear to 4=severe
Change from Baseline in weekly averaged Peak Pruritus Numerical Rating Scale (PP-NRS) at Week 16 | Baseline and Week 16
  The PP-NRS is a single item patient-reported outcome (PRO) measure assessing the worst itch in the last 24 hours. It will be assessed on a Numerical Rating Scale. The degree of itch will be scored on an 11-point scale, with 0 being "no itch" and 10 being the "worst itch imaginable."
Incidence of Treatment-Emergent (TE) Adverse Events (AE) | Up to Week 58
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A TEAE is defined as any AE with a start on or after the first administration of study intervention until 8 weeks after final administration.
Incidence of TE Serious Adverse Events (SAEs) | Up to Week 58
  An SAE is defined as any untoward medical occurrence that, at any dose, meets 1 or more of the criteria listed:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients or may require medical or surgical intervention to prevent any of the above.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 22733
Locations (7):
- United States (7):
  - Atd002 52015, Savannah, Georgia
  - Atd002 52017, Chicago, Illinois
  - Atd002 52012, New Albany, Indiana
  - Atd002 52001, Troy, Michigan
  - Atd002 52009, Troy, Michigan
  - Atd002 52010, Omaha, Nebraska
  - Atd002 52011, Frisco, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org